CLINICAL TRIAL: NCT05594277
Title: The Impact of Hospitalization After Major Surgery on Elderly Frail Patients: a Prospective Observational Study
Brief Title: Frailty and Surgery
Status: Completed | Type: Observational
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Francesca Moretto, Medical doctor, physician, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Other Study IDs: 421/CE
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgical elderly patients: Patients ≥ 70 years old, undergoing a major surgery in general and vascular surgery, urology, orthopedics at Maggiore della Carità University Hospital, Novara, Italy, having a General Practitioner listed in the Local Health Authority of Novara.

SUMMARY:
Frailty has been recently re-defined as a condition that is evident over time through an excess of vulnerability to stressors, with reduced ability to maintain or regain homeostasis after a destabilizing event, and occurrence of disability. Frailty has been often used to characterize the weakest and most vulnerable subset of older adults, because of age, comorbidities, social and emotional status leading to the lack of functional and psychological reserve and mining the capability to face acute events. Frail patients are becoming ever more present in Anesthesia and Intensive Care. In fact, 30 percent of surgery is conducted on patients ≥ 70 years old nowadays. It has been demonstrated that the impact of surgery and anesthesiologic risk are greater in older frail subjects, and that a low functional status is associated with increased mortality. Also, post-operative delirium and cognitive disfunction are more often seen in older patients. For this reason, the worsening of the global performance status, as functional status, mobility, and cognitive status may have a large impact on patient and caregivers' life. The primary objective is to evaluate the impact at three months after hospitalization following major surgery i.e., urology, general surgery, orthopedics, on the performance status as functional status, mobility, and cognitive status of patients ≥ 70 years old. Secondary objectives are to evaluate the necessity of domiciliary care assistance and re-hospitalization or rehabilitation center admissions in three months following surgery and to evaluate the impact of the type of anesthesia used in major surgery i.e., general vs regional anesthesia, on patient performance status.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years old
* Listed for major surgery in general and vascular surgery, urology, orthopedics
* Patient General Practitioner listed in the Local Health Authority of Novara

Exclusion Criteria:

* Barthel index at baseline < 16 in the activities of daily living section
* Barthel index at baseline < 11 in the mobility section
* Mini mental state examination at baseline < 11

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients affering to Maggiore della Carità University Hospital and Local Health Authority of Novara, Italy, listed for major surgery in general and vascular surgery, urology, orthopedics
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Worsening of the performance status as functional status, mobility, and cognitive status after hospitalization for major surgery | Three months
  Ten-point worsening of Barthel index globally, in the activities of daily living section and in the mobility section, and worsening of the mini mental state examination three months after surgery

SECONDARY OUTCOMES:
Necessity of domiciliary care assistance | Three months
  Necessity of domiciliary care assistance activation following hospital discharge after major surgery
Re-hospitalization or rehabilitation center admissions | Three months
  Necessity of re-hospitalization or rehabilitation center admissions in the three months after major surgery
Impact of the type of anesthesia used in major surgery, general vs regional anesthesia, on patient performance status | Three months
  Ten-point worsening of Barthel index globally, in the activities of daily living section and in the mobility section, and worsening of the mini mental state examination three months after surgery based on the type of anesthesia used in major surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Vaschetto, Professor, Study Chair — Università degli Studi del Piemonte Orientale Amedeo Avogadro
Locations (1):
- AOU Maggiore della Carità, Novara, Italy

REFERENCES:
- [Derived] Moretto F, Fracazzini M, Scotti L, Viarengo V, Gentilli S, Romito R, Volpe A, Leigheb M, Porta CM, Konrad P, Colombo D, Olivieri C, Della Corte F, Cammarota G, Vaschetto R. Major Elective Surgery Impact on Performance Status in Older Adults: A Prospective Observational Study. Health Sci Rep. 2025 Nov 2;8(11):e71438. doi: 10.1002/hsr2.71438. eCollection 2025 Nov. PMID 41189953